CLINICAL TRIAL: NCT05539027
Title: Efficacy of L-Ornithine L-Aspartate (LOLA) as an Adjunct to Branched Chain Amino Acids (BCAA) Enriched Solutions on Clinical Outcomes in ICU Patients With Hepatic Encephalopathy: a Randomized Controlled Trial
Brief Title: Efficacy of L-Ornithine L-Aspartate (LOLA) as an Adjunct to Branched Chain Amino Acids (BCAA) Enriched Solutions on Clinical Outcomes in ICU Patients With Hepatic Encephalopathy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ibrahim Mamdouh Esmat, Assistant Professor of Anesthesia and Intensive Care Department, Faculty of Medicine, Ain- shams University, Cairo, Egypt., Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FMASU MS 556/ 2022
Record Dates: First submitted 2022-09-07; First posted 2022-09-14 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Hepatic Encephalopathy
MeSH Terms: conditions — Hepatic Encephalopathy | interventions — Amino Acids, Branched-Chain; ornithylaspartate

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Treatment group) (Active Comparator)
  Interventions: Drug: Branched-chain amino acids (BCAA), enriched solution (Aminoleban) and L-ornithine L-aspartate (LOLA)
- Group 2 (Control group) (Active Comparator)
  Interventions: Drug: Branched-chain amino acids (BCAA), enriched solution (Aminoleban)

INTERVENTIONS:
Drug: Branched-chain amino acids (BCAA), enriched solution (Aminoleban) and L-ornithine L-aspartate (LOLA) — patients will receive branched-chain amino acids (BCAA), enriched solution (Aminoleban) and L-ornithine L-aspartate (LOLA)
  Arms: Group 1 (Treatment group)
Drug: Branched-chain amino acids (BCAA), enriched solution (Aminoleban) — patients will receive BCAA enriched solution (Aminoleban)
  Arms: Group 2 (Control group)

SUMMARY:
One of the most significant goals of hepatic encephalopathy (HE) treatment is to reduce ammonia levels by lowering its synthesis and enhancing its detoxification which can be achieved by using non-absorbable disaccharides, antibiotics, branched-chain amino acids (BCAA), L-ornithine L-aspartate (LOLA), and probiotics.

LOLA decreases ammonia, therefore, it is presumed to decrease agitated delirium in HE patients and thus decrease their need for other sedatives. On the other hand, BCAA improve mental function in HE patients by increasing the detoxification of ammonia in muscles.

DETAILED DESCRIPTION:
The most often utilized criteria for grading HE are the West Haven criteria (WHC). This grading distinguishes four levels of clinically evident hepatic encephalopathy.

West Haven criteria (WHC): [R]

Stage Consciousness

0. Normal

1. Mild lack of awareness
2. Lethargic
3. Somnolent but arousable
4. Coma

REFERENCES:

Ferenci P, Lockwood A, Mullen K, Tarter R, Weissenborn K, Blei AT. Hepatic encephalopathy-definition, nomenclature, diagnosis, and quantification: final report of the working party at the 11th World Congress of Gastroenterology, Vienna, 1998. Hepatology 2002; 35: 716-21.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Liver cirrhosis based on clinical, biochemical, radiological and/or histopathology.
* Patients having overt HE, West Haven criteria (WHC) grade III-IV.

Exclusion Criteria:

* Age < 21 years.
* Inability to obtain an informed consent from the first degree relative and/or legally authorized representative.
* Advanced cardiac or pulmonary disease.
* Presence of underlying chronic renal failure (serum creatinine > 3 mg/dL).
* Neurodegenerative disease (including head injury and drug intoxication).
* Major psychiatric illness.
* Use of sedatives or antidepressants.
* Pregnancy or breast-feeding .
* Hepatocellular carcinoma.
* Acute on top of chronic liver failure.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2022-09-20 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Reversal of Hepatic encephalopathy or change of Hepatic encephalopathy by two grades (according to West Havens Criteria) | 5 days of treatment
  Reversal of Hepatic encephalopathy or change of Hepatic encephalopathy by two grades (according to West Havens Criteria)

CONTACTS AND LOCATIONS:
Locations (1):
- Ain-Shams University Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided